CLINICAL TRIAL: NCT00187161
Title: Small Noncleaved Cell (SNCC), Non-Hodgkin Lymphoma (NHL), Large Cell NHL (B-Cell) and B-Cell Acute Lymphoblastic Leukemia (B-ALL) Study II
Brief Title: Treatment of Burkitt Lymphoma/Leukemia and B Large Cell NHL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: John T. Sandlund, MD / Principal Investigator, St. Jude Children's Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SJBCII
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Non-Hodgkin Lymphoma; Acute Lymphoblastic Leukemia, Mature B-Cell
Keywords: Mature B-Cell Leukemia; Non-Hodgkin Lymphoma; Burkitt's lymphoma; Small noncleaved cell non Hodgkin lymphoma; Large cell lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Vincristine; Cytarabine; Methotrexate; Etoposide; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Group A: Resected Stage I and resected abdominal Stage II
  Subjects will receive two courses (3 weeks apart) of COPAD.
  Interventions: Drug: Prednison, Vincristine, Cytarabine, Methotrexate, Etoposide, Cyclophosphamide, Doxorubicin
- B (Experimental): Group B: Other Stage II, Stage III, Stage IV or B-ALL M blast <70%; no CNS involvement.
  Subjects in Group B will receive one week of treatment of COP.
  Interventions: Drug: Prednison, Vincristine, Cytarabine, Methotrexate, Etoposide, Cyclophosphamide, Doxorubicin
- C (Experimental): Group C: B-ALL with >70% BM blasts; CNS involvement, Group B COP failures i.e., <20% reduction Treatment Pre-Induction
  Subjects will receive one week of treatment of COP.
  Interventions: Drug: Prednison, Vincristine, Cytarabine, Methotrexate, Etoposide, Cyclophosphamide, Doxorubicin

INTERVENTIONS:
Drug: Prednison, Vincristine, Cytarabine, Methotrexate, Etoposide, Cyclophosphamide, Doxorubicin — The additional information is contained in the Detailed Description section.

SUMMARY:
This is a pilot study to demonstrate that the modified LMB-89 treatment regimen for children with newly diagnosed small noncleaved cell NHL, large cell NHL (B-cell), and B-cell acute lymphoblastic leukemia can be delivered in this setting with acceptable toxicity.

DETAILED DESCRIPTION:
Group A: Resected Stage I and resected abdominal Stage II

Subjects will receive two courses (3 weeks apart) of COPAD as follows:

Cyclophosphamide (CTX) 500 mg/m2/day (divided q12 hrs) IV day 1, 2, 3 Vincristine (VCR) 2 mg/m2 (max 2.0 mg) IV day 1, 6 Prednisone 60 mg/m2/d (divided bid) PO day 1-5 Adriamycin 60 mg/m2 over 6 hrs IV day 1 GCSF 5 mcg/kg/day SQ will be given once a day starting on day 7 until blood counts recover.

Group B: Other Stage II, Stage III, Stage IV or B-ALL M blast <70%; no CNS involvement.

Treatment Pre-Induction

Subjects in Group B will receive one week of treatment of COP as follows:

CTX 300 mg/m2 IV day 1; VCR 1 mg/m2 (max 2.0 mg) IV day 1; Prednisone 60 mg/m2/day (divided bid) PO day 1-7; Methotrexate (MTX) and hydrocortisone (HC) into the spinal fluid (IT), each age adjusted, day 1; Induction -COPADM x 2 (COPAD M3 #1 (starting day 8 COP if greater than or equal to 20% reduction in tumor size by day 7 COP; if <20% then proceed to Group C starting at COPADM8 No. 1); COPADM3 #1 VCR 2 mg/m2 (max 2 mg) IV day 1; High-dose (HD) MTX 3 gm/m2 IV (over 3 hrs) day 1; MTX and HC each age adjusted IT day 2, 6 CTX 500 mg/m2/day (divided q12 hrs) IV day 2, 3, 4; Adriamycin 60 mg/m2 over 6 hrs IV; day 2; Prednisone 60 mg/m2 (divided bid) po day 1-5. G-CSF 5 mcg/kg/day starting day 7 until counts recover.

COPADM3 #2

Like COPADM #1 (above) except:

1. CTX - double dose (1 gm/m2/day) (divided q12 hr)
2. VCR - second dose given on day 6 Consolidation- CYM x 2 courses HDMTX 3 gm/m2 (over 3 hr) IV Day 1; MTX plus HC each age adjusted IT day 2; Cytarabine (Ara-C) 100 mg/m2/day CI/IV (x 5 days) day 2-6; Ara-C and HC each age adjusted IT day 7.

Maintenance Sequence 1 Prednisone 60 mg/m2/d (divided bid) PO day 1-5; HDMTX 3 gm/m2 (over 3 hr) IV Day 1; MTX plus HC each age adjusted IT day 2; CTX 500 mg/m2/day IV day 2, 3; Adriamycin 60 mg/m2 (over 6 hrs) IV day 3; VCR 2 mg/m2 (max 2 mg) IV day 1. G-CSF 5 mcg/kg/day starting day 6 until counts recover.

Group C: B-ALL with >70% BM blasts; CNS involvement, Group B COP failures i.e., <20% reduction Treatment Pre-Induction

Subjects will receive one week of treatment of COP as follows:

CTX 300 mg/m2 IV day 1 VCR 1 mg/m2 (max 2 mg) IV day 1 Prednisone 60 mg/m2/d (divided) bid po day 1-7 MTX + HC + Ara-C each age adjusted IT day 1, 3, 5 Leucovorin 15 mg/m2 q12 hr x 2 po day 2, 4 Induction-COPADM x 2

Subjects will begin induction therapy the day after COP is finished as follows:

COPADM8#1 VCR 2 mg/m2 (max 2 mg) IV day 1; HD MTX 8 gm/m2 (over 4 hrs) IV Day 1; MTX+HC+Ara-C each age adjusted IT day 1, 4, 6 (Ommaya, day 1); CTX 500 mg/m2/day divided every 12 hours IV day 2, 3, 4; Adriamycin 60 mg/m2 (over 6 hrs) IV day 2; Prednisone 60 mg/m2/day (divided bid) po/IV day 1-5. G-CSF 5 mcg/kg/day starting day 7 until counts recover.

COPADM8 #2

Like COPAD M8 #1 except:

1. CTX-double dose (1 gm/m2/day) (divided q12hs) IV
2. VCR - 2nd dose given on day 6 Consolidation - CYVE x 2 courses Ara-C 50 mg/m2/12 hrs CI/IV Day 1-5; HD Ara-C 3 gm/m2/day IV over 3 hours Day 2-5; VP-16 200 mg/m2/day IV over 2 hours Day 2-5.

Maintenance: Subjects will receive four courses of chemotherapy during continuation. Each course will use different chemotherapy drugs.

Sequence 1 Prednisone 60 mg/m2/day (divided bid) po/IV day 1-5; HD MTX 8 gm/m2 (over 4 hrs) IV Day 1; MTX+HC+Ara-C each age adjusted IT day 2 (Ommaya, day 2) CTX 500 mg/m2 IV day 2, 3; Adriamycin 60 mg/m2 (over 6 hrs) IV day 3; VCR 2 mg/m2 (max 2 mg) IV day 1. G-CSF 5 mcg/kg/day starting day 7 until counts recover.

Sequence 2 Ara-C 100 mg/m2/day (divided q12 hrs) SQ Day 1-5; VP-16 150 mg/m2/day (over 2 hrs) IV Days 1-3; G-CSF 5 micro g/kg SQ Days 6 until counts recovery; MTX+HC+Ara-C each age adjusted IT Day 1 (CNS positive, only) Ommaya Day 1 (CNS positive, only) Sequence 3 Prednisone 60 mg/m2/day (divided bid) po day 1-5; CTX 500 mg/m2/day IV day 1, 2; Adriamycin 60 mg/m2 (over 6 hrs) IV day 2; VCR 2 mg/m2 (max 2 mg) IV day 1; G-CSF 5 mcg/kg SQ starting day 6 until counts recover; MTX+HC+Ara-C each age adjusted IT Day 1 (CNS positive, only) Ommaya Day 1 (CNS positive, only).

Sequence 4 Ara-C 100 mg/m2/day (divided q12 hrs) SQ Day 1-5; VP-16 150 mg/m2/day (over 2 hrs) IV Days 1-3; G-CSF 5 mcg/kg SQ days 6 until counts recover; MTX+HC+Ara-C each age adjusted IT Day 1 (CNS positive, only) Ommaya Day 1 (CNS positive, only)

Intrathecal (IT) Treatment doses and volume are as follows:

< than 1 year, MTX 8 mg, HC 8 mg, Ara C 15 mg, Volume 8 ml; Age 12-23 mo, MTX 10 mg, HC 10 mg, Ara C 20 mg, Volume 10 ml; Age 24-35 mo, MTX 12 mg, HC 12 mg, Ara C 25 mg, Volume 12 ml; Age ≥3 yr, MTX 15 mg, HC 15 mg, Ara C 30 mg. Volume 15 ml Ommaya Reservoir Treatment (CNS positive only) Age ≥3 yr, MTX 6 mg, HC 15 mg, Ara C 50 mg/m2 (50 mg max) Volume 3 ml

ELIGIBILITY:
Inclusion Criteria:

* Subject must be previously untreated, except for steroids.
* Subject must be less than or equal to 18 years of age.
* Subject must have a histologic diagnosis of small noncleaved cell (SNCC) NHL or large cell NHL (B-cell), or B-cell acute lymphocytic leukemia.

Exclusion Criteria:

* Previously treated disease

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 1994-11; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The purpose of this study is estimate the complete response, event-free survival, and overall survival in patients with small non-cleaved cell non-Hodgkin lymphoma or large cell NHL, or Burkitt leukemia/B-cell ALL treated with a modified LMP-89 regimen. | 8-9 years

CONTACTS AND LOCATIONS:
Overall Officials: John T. Sandlund, M.D., Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org